CLINICAL TRIAL: NCT03052946
Title: A Prospective Randomized Study Between the Use of Bulking Agent and the Endoanal Electrostimulation Therapy in Patients With Mild or Moderate Anal Incontinence
Brief Title: Bulking Agent Versus Electrostimulation Therapy in Anal Incontinence
Acronym: Bulking
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Leonardo Alfonso Bustamante, Surgeon research at the colon and rectum service. Gastroenterology Department, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09082009
Record Dates: First submitted 2017-02-10; First posted 2017-02-14 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Fecal Incontinence
Keywords: fecal incontinence, anorectal manometry, bulking agents
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Intervention Model Description: Bulking agents
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bulking agent (Active Comparator): Bulking agent in fecal incontinence
  Interventions: Procedure: Bulking agent
- Endoanal electrostimulation (Placebo Comparator): Endoanal electrostimulation in fecal incontinence
  Interventions: Procedure: Endoanal electrostimulation

INTERVENTIONS:
Procedure: Bulking agent — Filling bulking agent in the anal canal
  Arms: Bulking agent
Procedure: Endoanal electrostimulation — The technique used will be with a frequency of 30 to 40 Hz with pulse width of 200 ms with maximum intensity of 800mAmp and duration of 30 minutes
  Arms: Endoanal electrostimulation

SUMMARY:
Randomized trial with a estimated number of 60 patients with mild or moderate anal incontinence at the clinic Physiology of the Hospital das Clínicas of the Medical School of the University of São Paulo (HC-FMUSP).

* Exclusion criteria: symptoms of anal incontinence for less than six months, with severe anal incontinence, associated external anal sphincter damage, past pelvic radiotherapy, evidence of perineal sepsis, rectal prolapse, anorectal cancer, inflammatory bowel disease, malignant disease Congenital formation, scleroderma, Parkinson's disease, immunosuppression and ongoing gestation. In addition, those patients who do not agree to participate in the survey will be excluded.
* The study will have 4 phases: preoperative, surgical, recent postoperative and later postoperative

DETAILED DESCRIPTION:
* Prospective randomized trial
* Estimated number of 60 patients with mild or moderate anal incontinence with isolated anal sphincter muscle damage or evidence of anal incontinence without verification of anatomical damage to the anorectal sphincter complex with dysfunction or inadequate action of the internal anal sphincter accompanied at the outpatient clinic Physiology of the Hospital das Clínicas of the Medical School of the University of São Paulo (HC-FMUSP).
* Exclusion criteria: symptoms of anal incontinence for less than six months, with severe anal incontinence, associated external anal sphincter damage, past pelvic radiotherapy, evidence of perineal sepsis, rectal prolapse, anorectal cancer, inflammatory bowel disease, malignant disease Congenital formation, scleroderma, Parkinson's disease, immunosuppression and ongoing gestation. In addition, those patients who do not agree to participate in the survey will be excluded.
* The study will have 4 phases: preoperative, surgical, recent postoperative and later postoperative

ELIGIBILITY:
Inclusion Criteria:

* Moderate fecal incontinence

Exclusion Criteria:

* Severe fecal incontinence
* Pelvic radiotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-02-28 (Estimated); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Fecal incontinence | 6 months
  Score of Fecal Incontinence

IPD SHARING:
Plan to Share IPD: No